CLINICAL TRIAL: NCT02249936
Title: A Phase 1, Single-Center, Randomized, 3-Way Cross-Over, Open Label Study to Evaluate the Pharmacodynamics of Different Formulations of AZD1722 in Healthy Volunteers Taking Omeprazole
Brief Title: A Phase 1 Study to Examine the Pharmacodynamics of Different AZD1722 Formulations
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ardelyx (Industry)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D5611C00002
Record Dates: First submitted 2014-09-24; First posted 2014-09-26 (Estimated); Last update posted 2014-09-26 (Estimated); Status verified 2014-09

CONDITIONS: Healthy
Keywords: Volunteers
MeSH Terms: interventions — tenapanor; Omeprazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- AZD1722 HCl Capsule (Experimental): 15 mg bid AZD1722 HCl and 20 mg bid Omeprazole
  Interventions: Drug: AZD1722; Drug: Omeprazole
- AZD1722 HCl Tablet (Experimental): 15 mg bid AZD1722 HCl and 20 mg bid Omeprazole
  Interventions: Drug: AZD1722; Drug: Omeprazole
- AZD1722 Free-base Tablet (Experimental): 15 mg bid AZD1722 and 20 mg bid Omeprazole
  Interventions: Drug: AZD1722; Drug: Omeprazole

INTERVENTIONS:
Drug: AZD1722
  Other Names: Tenapanor; RDX5791
Drug: Omeprazole

SUMMARY:
The study is designed to evaluate safety, tolerability, pharmacodynamics and pharmacokinetics of different formulations of AZD1722 in healthy male and female subjects taking Omeprazole.

ELIGIBILITY:
Inclusion Criteria:

* Healthy man or woman
* Body mass index between 18 and 29.9 kg/m2

Exclusion Criteria:

* Diagnosis or treatment of any clinically symptomatic biochemical or structural abnormality of the gastrointestinal (GI) tract
* Any surgery on the small intestine or colon, excluding appendectomy or cholecystectomy or any other condition known to interfere with absorption, distribution, metabolism or excretion of drugs
* Clinical evidence of significant cardiovascular, respiratory, renal, hepatic, gastrointestinal, hematologic, metabolic, endocrine, neurologic, psychiatric disease, or any condition that may interfere with the subject successfully completing the trial or that would present a safety risk

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2013-02; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Number of patients with adverse events | 8 days
  Measurement of safety laboratories, ECGs, vitals signs and physical exams

SECONDARY OUTCOMES:
Sodium levels in stool and urine | 8 days
  Pharmacodynamic activity
Plasma drug concentration to calculate AUC | 8 days
  Pharmacokinetics

CONTACTS AND LOCATIONS:
Overall Officials: David P Rosenbaum, Ph.D., Study Director — Ardelyx, Inc
Locations (1):
- ICON Development Solutions, Omaha, Nebraska, United States